CLINICAL TRIAL: NCT02791360
Title: Evaluation of Anatomy, Clinical and Neuropsychological Long-term Sequelae of Patients Treated With Radiation Therapy for Brain Tumor
Acronym: TCSEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TCSEQ
Record Dates: First submitted 2016-05-17; First posted 2016-06-06 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Brain Neoplasms
Keywords: Brain; Radiotherapy; MRI; Sequelae
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI evaluation (Other): Patient pretreated for brain tumor and witness
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI

SUMMARY:
Through this study, the investigators believe to describe more accurately the damage caused by brain radiation therapy in the long term.

ELIGIBILITY:
Inclusion Criteria:

In the case group:

* A history of solid brain tumor or haematological histologically proven.
* Patients previously treated with radiotherapy in this brain tumor (greater than or equal to 36 Gy dose).
* Radiotherapy treatment on a tumor in place or operated.
* Decline at least 10 years from the end of radiotherapy.
* Treatment with isocentric conformal radiotherapy.
* No other radiation therapy for locally recurrent brain metastases or new brain tumor.
* Lack of known brain metastases or meningeal carcinomatosis.

For the control group:

* Patients previously treated for cancer and disease relapse free for 10 years.
* No brain radiotherapy treatment.
* Lack of treatment with anti-cancer chemotherapy.
* Women of childbearing potential must be under effective contraception.
* Pairing according to age, sex, arms director and socio-cultural level.

For two groups:

* Man or woman aged (e) of minimum 18 years.
* Topic fluent French and comprising well.
* Free and Informed Consent signed.
* The subject should be affiliated to an appropriate social security system
* No cons-indication to MRI.
* The subject must have at least one primary school level

Exclusion Criteria:

In the case group:

* Brain radiotherapy carried out by intensity modulation technique.
* Radiation dose less than 36 Gy on the brain.
* Subject with against-indication to MRI.

For the control group:

* Previous history of brain radiotherapy.
* Previous history of brain surgery.
* Central neurological disorders, such as seizures, uncontrolled.

For two groups:

* Current Topics in oral chemotherapy or intravenous.
* Subject pregnant.
* Subject is not fluent in French or including bad.
* Any geographical conditions, social or associated psychopathology that could compromise the patient's ability to participate in the study.
* Participation in a therapeutic trial for less than 30 days.
* A person not affiliated with a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patient with MRI abnormality | up to 4 weeks
  To evaluate the proportion of patients with at least one abnormality on an imaging test

SECONDARY OUTCOMES:
MRI diffusion abnormality | up to 4 weeks
MRI perfusion abnormality | up to 4 weeks
MRI vascular morphologic abnormalities | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France